CLINICAL TRIAL: NCT02011503
Title: A Randomized Controlled Clinical Trial Evaluating The Application Of Dehydrated Human Amnion/ Chorion Membrane (dHACM) Plus Standard Of Care Vs. Standard Of Care Alone In The Treatment Of Venous Leg Ulcers
Brief Title: Use of dHACM in the Treatment of Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFVLU003
Record Dates: First submitted 2013-11-21; First posted 2013-12-13 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dHACM (Experimental): Application of multi-layer compression therapy with application of dHACM.
  Interventions: Procedure: Multi-layer compression therapy; Other: Application of dHACM
- Control (Other): Application of multi-layer compression therapy without application of dHACM.
  Interventions: Procedure: Multi-layer compression therapy

INTERVENTIONS:
Procedure: Multi-layer compression therapy — Application of multi-layer compression therapy.
Other: Application of dHACM — Application of dHACM to ulcer.
  Arms: dHACM

SUMMARY:
The overall objective of this study is to evaluate the effectiveness of dehydrated human amnion/ chorion membrane (dHACM) in reducing time to complete wound closure in patients with venous leg ulcers (VLUs).

ELIGIBILITY:
Inclusion Criteria:

1. Index ulcer characteristics:

   1. Full-thickness venous leg ulcer for ≥ 30 days
   2. Ulcer area after debridement is ≥ 1 cm² and ≤ 25 cm² at the randomization visit
   3. Has a clean, granulating base with minimal adherent slough
2. Subject has completed 14 day run-in period with ≤ 25% wound area reduction post-debridement.
3. Have one of the following:

   * Ankle Brachial Pressure Index (ABI) > 0.75. (Calculations will be made using measurements from both posterior tibial and dorsalis pedis arteries as well as both arms) OR
   * Have venous insufficiency confirmed by duplex ultrasound examination for valvular or venous incompetence.
4. Age ≥ 18.
5. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
6. Ability to read/understand and sign Informed Consent and Release of Medical Information Forms.
7. Ability to understand and comply with weekly visits and follow-up regimen.

Exclusion Criteria:

1. Index Ulcer Assessment - Index ulcer meeting the following criteria will not be eligible for enrollment:

   1. Penetrates down to muscle, tendon, or bone
   2. Presence of another venous ulcer ≤ 2 cm from index ulcer
   3. Is deemed by the Investigator to be caused by a medical condition other than venous insufficiency
   4. Exhibits clinical signs and symptoms of infection
   5. If in the opinion of the Investigator, the wound is suspicious for cancer, the subject should undergo an ulcer biopsy to rule out carcinoma. If carcinoma is ruled out, the subject may be re-screened.
   6. Located on the dorsum of the foot or with more than 50% of the ulcer below the malleolus
2. Prior therapies - Subjects receiving treatment with any of the following will not be eligible for enrollment:

   1. In the last 7 days - Negative pressure wound therapy of the index ulcer
   2. In the last 7 days - Hyperbaric oxygen therapy
   3. In the last 30 days - Treatment with cytotoxic chemotherapy, application of topical steroids to the ulcer surface, or use of ≥ 14 days of immune-suppressants (including systemic corticosteroids); or, subject is anticipated to require such medications during the course of the study
   4. In the last 30 days - study ulcer treatment with any advanced therapy, including EpiFix®, tissue engineered materials (e.g. Apligraf® or Dermagraft®), or other scaffold materials (e.g. OASIS® Wound Matrix, MatriStem® Wound Matrix)
   5. In the last 30 days - Subject has been on any investigational drug(s) or therapeutic device(s)
   6. In the last 8 weeks - Amputation or revascularization (surgical or stenting) to the affected leg
   7. Any history of radiation at the ulcer site
   8. Any prior participation in a MiMedx® study
   9. Study ulcer has undergone ≥ 12 months of continuous high strength compression therapy over its duration
3. Subject criteria that will make subject ineligible for enrollment:

   1. Known osteomyelitis or active cellulitis at wound site
   2. Hemoglobin A1C >12 in the last 60 days prior to randomization
   3. Active malignant disease or subject is less than 1 year disease-free
   4. NYHA Class III and IV congestive heart failure (CHF), as defined by the following criteria: Class III: Symptoms with moderate exertion; Class IV: Symptoms at rest
   5. Auto-immune disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS) or HIV
   6. Allergy or known sensitivity to Aminoglycosides such as gentamicin sulfate and/or streptomycin sulfate
   7. Known allergy to the components of the multi-layer compression bandaging, or who cannot tolerate MLCT
   8. Presence of any condition (including current drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol in the judgment of the Investigator
   9. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08-05 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Time to 100% epithelialization of study ulcer | 12 weeks

SECONDARY OUTCOMES:
Proportion of patients in both groups with complete wound healing at 12 weeks | 12 weeks

OTHER OUTCOMES:
Comparison of Quality of Life as assessed by Short Form 36 (SF-36) | 16 weeks
Crossover Subject Analysis | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Don Fetterolf, MD, Study Director — MiMedx Group, Inc.
Locations (15):
- United States (15):
  - Associated Foot & Ankle Specialists, PC, Phoenix, Arizona
  - ILD Research, Carlsbad, California
  - Center for Clinical Research, Inc., Castro Valley, California
  - Center for Clinical Research, Inc., Fair Oaks, California
  - Limb Preservation Platform, Inc., Fresno, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - VA Northern California, Mather, California
  - Center for Clinical Research, Inc., San Francisco, California
  - Atlanta Veteran's Administration, Decatur, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - VA Western New York Health Care System, Buffalo, New York
  - Center for Clinical Research, Inc., Eugene, Oregon
  - SGM Physicians, Haverford, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - William Jennings Bryan Dorn Veterans Affairs Medical Center, Columbia, South Carolina